CLINICAL TRIAL: NCT00604734
Title: A Prospective Clinical Study On A Total Hip Resurfacing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EU-8
Record Dates: First submitted 2007-12-23; First posted 2008-01-30 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Arthritis; Avascular Necrosis
MeSH Terms: conditions — Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ReCap (Other): ReCap Total Hip Resurfacing System
  Interventions: Device: ReCap Total Hip Resurfacing System

INTERVENTIONS:
Device: ReCap Total Hip Resurfacing System — This is a hip resurfacing system.
  Other Names: Total hip resurfacing; ReCap

SUMMARY:
This prospective clinical study is to demonstrate the efficacy and safety of ReCap Total Hip Resurfacing System.

DETAILED DESCRIPTION:
The study is designed as a prospective, multi-center, non-randomized study. It is designed to evaluate the effects of metal-on-metal acetabular articulating bearing surfaces.

The device will be used in conjunction with a cemented metal femoral resurfacing prosthesis.

The objective of this clinical investigation is to evaluate the safety and effectiveness of the metal-on-metal Recap Total Resurfacing System.

Performance will be assessed trough Harris Hip Score, radiographic evaluation at various postoperative visits. Adverse events and revisions will be documented for safety assessments.

Primary endpoints:

* Total Harris hip score
* Device revisions or removals

Secondary endpoints:

* Total Harris hip score
* Radiographic changes as evidenced by:

I. Acetabular component migration, change in angle of inclination or presence of osteolysis II. Femoral component subsidence, femoral neck Fracture or presence of osteolysis

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a preoperative Total Harris Hip Score of < 70
2. Conservative treatment has proven unsuccessful
3. Primary hip surgery
4. Patients requiring hip resurfacing for degenerative joint disease (inflammatory or non- inflammatory) or any of the composite diagnoses of:

   1. Osteoarthritis
   2. Avascular necrosis
   3. Legg Perthes
   4. Rheumatoid Arthritis
   5. Juvenile Rheumatoid Arthritis
   6. Systemic Lupus Erythematosus
   7. Developmental Dysplasia, which does not prevent stable acetabular reconstruction
   8. Post traumatic arthritis S. Patients at least 18 years of age

6. Patients of all races and gender 7. Patients who are able to follow post-operative care instructions 8. Patients who are willing and able to return for scheduled follow-up evaluations 9. Patient has signed the IRB approved Informed Consent Form

Exclusion Criteria:

1. Patients with a preoperative Total Harris Hip Score of > 70
2. Previous prosthetic hip replacement device (including other surface arthroplasty, endoprosthesis,etc) in the operative hip
3. Contralateral hip prosthesis (total hip replacement or surface replacement),including staged or simultaneous procedures
4. Developmental dysplasla, which prevents stable acetabular reconstruction
5. Patients with previous Girdlestone procedures
6. Patients with above knee amputation of the contralateral and/or ipsilateral leg
7. Severe osteoarthritis or marked bone loss,which would preclude proper fixation of the prosthetic device(s)
8. Active or suspected systemic or localized Infection
9. Parkinson's or Alzheimer's Disease
10. Patients with severe instability or deformity of the ligaments and/or surrounding soft tissue,which would preclude stability of the prosthesis
11. Patients less than 18 years of age
12. Patients with condition(s) that may Interfere with the survival of the femoral resurfacing or acetabular replacements or their outcomes,including Paget's Disease, Charcot's Disease, Sickle Cell Anemia or traits Severe osteoporosis compromising bone stock (I.e.Dorr type C bone Lower extremity muscular atrophy Neuromuscular disease
13. Patients with a clinical conditions that may limit follow-up,including: immunocompromised conditions, hepatitis, active tuberculosis, neoplastic disease, chronic renal failure, organ transplant recipients, known terminal disease process
14. Patients with a "fused"hip
15. Patients with metal allergy or hypersensitivity
16. Participation in a study of any investigational product (drug or device) within the past 12 months
17. Prisoners,known drug or alcohol abuser,or mentally incompetent individuals
18. Systemic steroids within 6 months
19. Patients with a known malignancy
20. Patients who are pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2004-10; Primary Completion 2007-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score, Device Revision/Removal, Radiographic Evaluation | 2 years postoperative

SECONDARY OUTCOMES:
Complications | Anytime

CONTACTS AND LOCATIONS:
Overall Officials: Jo De Schepper, MD, Principal Investigator — AZ Nikolaas
Locations (1):
- Az Nikolaas Campus Sint Niklaas, Sint-Niklaas, Belgium